CLINICAL TRIAL: NCT05746260
Title: Investigating Consolidation of Motor Learning in the Context of Recovery After Stroke
Brief Title: Sleep and Motor Learning in Stroke
Acronym: SMiLES
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: PID 16062
Record Dates: First submitted 2023-02-17; First posted 2023-02-27 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Stroke
Keywords: Rehabilitation; Motor Consolidation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will explore whether sleep disruption in the sub-acute phase of stroke explains variation in clinical motor outcomes, and whether this relationship is mediated by variation in behavioural measures of overnight consolidation.

DETAILED DESCRIPTION:
Rehabilitation of movement after stroke depends on motor learning. Motor learning involves not only improvement during practice but also improvement between sessions, known as consolidation of learning. Consolidation of learning depends on good sleep quality. However, there is growing evidence that sleep is disrupted after stroke, and it was recently shown that patients with poorer sleep show slower recovery of function and worse motor outcomes. This might occur because sleep disruption impairs consolidation directly or might reflect other factors that influence both sleep and clinical outcomes. This study aims to test whether the relationship between sleep disruption and clinical outcomes after stroke depends on consolidation of motor learning.

In people with stroke affecting the upper limb, the investigators will (1) test whether sleep measures in the sub-acute phase explains variation in clinical motor outcomes, taking into account recovery potential (as per the PREP2 algorithm(Predict REcovery Potential; www.presto.auckland.ac.nz)), demographic factors (age and sex) and other covariates as required (e.g. stroke severity, presence of sleep disorders, mood, physical activity), and (2) test whether this relationship is mediated by variation in behavioural measures of overnight motor consolidation.

The design is a longitudinal observational study. Participants will be recruited within 1 month of stroke onset from stroke wards. At baseline (≤ 1 month post-stroke), the investigators will use the PREP2 algorithm (www.presto.auckland.ac.nz) to ascertain expected upper limb recovery potential. This involves an assessment of arm movement and, for some participants, Transcranial Magnetic Stimulation to assess corticospinal tract integrity. The investigators will also record participant demographics, stroke severity (National Institute for Health Stroke Scale; NIHSS), and medications.

At approximately 1 month post-stroke the investigators will obtain sleep measures (actigraphy, electroencephalography, and questionnaires), assess mood (questionnaire) and test for motor consolidation (using an upper limb motor learning task). The investigators will also record medications, stroke severity (modified Rankin Scale questionnaire), and assess the possible presence of sleep disorders (sleep screening questionnaires), physical activity (actigraphy). The investigators will collect information about how much, if any, motor rehabilitation and sleep therapy the participants have received (questionnaire).

At 6 months post-stroke the investigators will obtain sleep measures (actigraphy, and questionnaire) and assess motor outcomes (upper limb ability, whole body motor impairment, hand dexterity, and mobility). The investigators will also record medications and assess mood (questionnaire), stroke severity (modified Rankin Scale questionnaire), physical activity (actigraphy), and information about how much, if any, motor rehabilitation and sleep therapy the participants have had (questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study OR a positive opinion from a consultee is provided by a family member or carer (relative or friend) willing to provide personal consultee (PC) advice
* Aged 18 years or above
* Within 1 month of onset of stroke affecting the upper limb as confirmed by clinical diagnosis

Exclusion Criteria:

* Other neurological condition affecting movement (such as Parkinson's disease, Multiple Sclerosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with stroke affecting the upper limb
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Sleep fragmentation at 1-month | 1 month post-stroke
  Assessed using actigraphy (wearable activity monitor) over 7-nights (more fragmentation indicates worse sleep).
Symptoms of insomnia at 1-month | 1 month post-stroke
  Assessed using the Sleep Condition Indicator, a questionnaire assessing self-reported insomnia symptoms (range 0-32, higher scores indicate fewer symptoms of insomnia)
Upper limb ability | 6 month post-stroke
  Assessed using the Action Research Arm Test (range 0-57, higher score indicates better upper limb ability)
Behavioural motor consolidation | 1 month post-stroke
  Assessed as change in motor performance on a sequential button pressing task (movement time, in seconds) from training to retest

SECONDARY OUTCOMES:
Whole body motor impairment | 6 months post-stroke
  Assessed using the Fugl-Meyer Assessment, range 0-100 (higher score indicates better functional mobility)
Hand dexterity | 6 months post-stroke
  Assessed using the Nine Hole Peg Test, scored as the number of pegs placed in 30 seconds (greater number of pegs indicates better hand dexterity)
Mobility | 6 months post-stroke
  Assessed using the Rivermead Mobility Index, range 0-15 (higher score indicates better functional mobility)
Estimated Total Sleep Time | 1 and 6 months post-stroke
  Assessed using actigraphy (wearable activity monitor) over 7-nights
Wake After Sleep Onset | 1 and 6 months post-stroke
  Assessed using actigraphy (wearable activity monitor) over 7-nights (higher amount of wake after sleep onset indicates worse sleep)
Symptoms of insomnia at 6-months | 6 months post-stroke
  Assessed using the Sleep Condition Indicator, a questionnaire assessing self-reported insomnia symptoms (range 0-32, higher scores indicate fewer symptoms of insomnia)

OTHER OUTCOMES:
Electroencephalography (EEG) Sleep Measures | 1 month post-stroke
  At home electroencephalography (EEG) headband for assessing sleep measures (e.g. sleep spindle amplitude, spindle density, sleep staging, cross-frequency coupling)
Mood (Depression) | 1 and 6 months post-stroke
  Assessed using the Patient Health Questionnaire (8-item), range 0-24 (higher values indicate more depressive symptoms)
Risk of Obstructive Sleep Apnoea | 1 month post-stroke
  Assessed using the STOP BANG questionnaire, range 0-8 (higher values indicate higher risk)
Presence of Sleep Disorders | 1 month post-stroke
  Assessed using the Sleep Disorders Screening questionnaire. Positive responses within sub-groups of questions indicate potential presence of specific sleep disorders.
Stroke severity | 1 and 6 months post-stroke
  Assessed using the modified Rankin Scale, range 0-6 (higher values indicate more severe stroke)
Stroke severity | Baseline
  Assessed using the National Institute for Health Stroke Scale (NIHSS), range 0-42 (higher values indicate greater severity)
Physical activity | 1 and 6 months post-stroke
  Assessed using actigraphy (wearable activity monitor) over 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Johansen-Berg, Professor, Principal Investigator — University of Oxford
Locations (1):
- Wellcome Centre for Integrative Neuroimaging (WIN), Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified data are available upon reasonable request
Supporting Information: Study Protocol
Time Frame: Following publication of results
Access Criteria: Available upon reasonable request

REFERENCES:
- [Derived] Weightman M, Robinson B, Mitchell MP, Garratt E, Teal R, Rudgewick-Brown A, Demeyere N, Fleming MK, Johansen-Berg H. Sleep and motor learning in stroke (SMiLES): a longitudinal study investigating sleep-dependent consolidation of motor sequence learning in the context of recovery after stroke. BMJ Open. 2024 Feb 13;14(2):e077442. doi: 10.1136/bmjopen-2023-077442. PMID 38355178